CLINICAL TRIAL: NCT01892423
Title: Daily Advance Cetaphil Moisturizing Lotion: Human Repeat Insult Patch Test
Brief Title: Repeat Insult Patch Test for Daily Advance Cetaphil Moisturizing Lotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04SPR.US10044
Record Dates: First submitted 2013-06-26; First posted 2013-07-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2013-06

CONDITIONS: Skin Irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetaphil Moisturizing Lotion Daily Advance (Experimental): Each subject had Cetaphil Moisturizing Lotion Daily Advance applied
  Interventions: Other: Cetaphil Moisturizing Lotion Daily Advance

INTERVENTIONS:
Other: Cetaphil Moisturizing Lotion Daily Advance

SUMMARY:
Human repeat insult patch test to assess the potential for Cetaphil Moisturizing Lotion Daily Advance to induce sensitization to the skin

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Good health
* willingness to cooperate and participate
* willingness to avoid topical products at test sites
* willingness to avoid direct sun exposure to test sites

Exclusion Criteria:

* Individuals with active psoriasis or eczema
* individuals with sunburn, acne, abrasions, scar tissue, or tattoos on test sites, or disease of skin that might interfere
* individuals who have had a mastectomy with axillary nodes were removed
* individuals receiving anticancer, immunosuppressive treatments or medications, or radiation
* pregnant, nursing, or planned to become pregnant
* use of topical steroids or drugs at test sites
* active or untreated skin cancer
* active hepatitis
* current routine or frequent use of high doses of anti-inflammatory drugs
* individuals who have had les than two week rest period since completion of previous patch testing on upper back or upper arms
* individuals with uncontrolled metabolic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Irritation responses | average of 5 weeks
  all patients will be assessed at 14 visits for redness (erythema), spreading, weeping, papules, vesicles, and bullae at application site

CONTACTS AND LOCATIONS:
Overall Officials: James H Herndon, MD, FAAD, Principal Investigator
Locations (1):
- Thomas J Stephens and Associates Inc, Carrollton, Texas, United States